CLINICAL TRIAL: NCT01104233
Title: Pain Outcomes Following Video-Assisted Thoracic Surgery (VATS) With Rigid Spreading Versus Soft Spreading (Using LAP Protector)
Brief Title: Pain Outcomes Following Video-Assisted Thoracic Surgery (VATS) With LAP Protector
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: The First Affiliated Hospital of Guangzhou Medical College, Guangzhou Medical College
Other Study IDs: FAHG20100320
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Last update posted 2010-04-15 (Estimated); Status verified 2010-03

CONDITIONS: Lung Cancer
Keywords: Video-assisted Thoracoscopic Surgery; Soft spreading; LAP Protector
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- The soft spreading: Patients with lung cancer underwent Video-assisted Thoracoscopic Surgery (VATS) with soft spreading (using LAP Protector).
  Interventions: Device: LAP Protector
- The rigid spreading: Patients with lung cancer underwent Video-assisted Thoracoscopic Surgery (VATS) with rigid spreading.

INTERVENTIONS:
Device: LAP Protector — The LAP Protector is a device that consists of two flexible rings made of superelasticity alloys covered with polyurethane polyamide, and a thin silicone rubber membrane that is attached to the outer rim of the two rings
  Groups: The soft spreading

SUMMARY:
The purpose of this study is to see if different types of spreading (rigid or soft) of Video-assisted Thoracoscopic Surgery (VATS) for lung cancer have different effects on pain.

DETAILED DESCRIPTION:
The Lap-Protector (Hakko Co., Japan) is a device that consists of two flexible rings made of superelasticity alloys covered with polyurethane polyamide, and a thin silicone rubber membrane that is attached to the outer rim of the two rings. If the two rings are pulled apart, the device assumes a cylindrical shape. The outer diameter of each flexible ring is 12 cm, and this device can be used for minilaparotomy wounds between 5 and 9cm long.

ELIGIBILITY:
Inclusion Criteria:

* Non-small cell lung cancer stage IB - IIIA
* ECOG status 0-1

Exclusion Criteria:

* Prior chemotherapy and/or radiation therapy for lung cancer
* Peripheral neuropathy > grade 1
* Concurrent other malignancies, other than basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* Medical condition that will not permit treatment or follow up according to the protocol
* Pregnant or nursing women
* HIV-positive patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-small cell lung cancer
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-10 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Compare the level of postoperative pain between the rigid and soft spreading groups | 1 day
  The level of postoperative pain was measured by Visual Analogue Scale (VAS).

SECONDARY OUTCOMES:
Compare early postoperative analgesic requirements between the rigid and soft spreading groups | 1 week
  Postoperative analgesic requirements (e.g. the amount of morphine titration).

CONTACTS AND LOCATIONS:
Overall Officials: Jianxing He, MD, FACS, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical College, Guangzhou, Guangdong, China